CLINICAL TRIAL: NCT07195487
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Center Clinical Study to Assess the Safety, Efficacy, and In-Use Tolerability of a Fermented Hair Growth and Scalp Health Serum in Subjects With Mild to Moderate Hair Thinning.
Brief Title: A Clinical Study to Evaluate the Safety, Effectiveness and In-Use Tolerability of Hair Growth and Scalp Health Serum in Subjects With Mild to Moderate Hair Thinning.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Blossom Microbiotics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB250022-BM_1.0_10Sep25
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Thinning Hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Extract Hair Growth and Scalp Health Serum (Experimental): Mode of Usage: Apply the serum directly to the scalp using the rollerball applicator. Gently roll the ball over thinning or affected areas of the scalp. Gently massage the serum into the scalp with clean fingertips to help it absorb fully. Ensure liquid is visible on the scalp and reapply until you feel a cooling wet sensation during application - this confirms the mechanism is working and that a good amount of product is being delivered.
  Frequency: Apply the treatment twice daily- once after morning shower and once before bed time. immediately after shower and at night before bed.
  Route of administration: Topical Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Interventions: Other: Fermented Extract Hair Growth and Scalp Health Serum
- Placebo Hair Growth and Scalp Health Serum (Placebo Comparator): Mode of Usage: Apply the serum directly to the scalp using the rollerball applicator. Gently roll the ball over thinning or affected areas of the scalp. Gently massage the serum into the scalp with clean fingertips to help it absorb fully. Ensure liquid is visible on the scalp and reapply until you feel a cooling wet sensation during application - this confirms the mechanism is working and that a good amount of product is being delivered.
  Frequency: Apply the treatment twice daily - once after morning shower and once before bed time. immediately after shower and at night before bed.
  Route of administration: Topical Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight
  Interventions: Other: Placebo Hair Growth and Scalp Health Serum

INTERVENTIONS:
Other: Fermented Extract Hair Growth and Scalp Health Serum — Mode of Usage: Apply the serum directly to the scalp using the rollerball applicator. Gently roll the ball over thinning or affected areas of the scalp. Gently massage the serum into the scalp with clean fingertips to help it absorb fully. Ensure liquid is visible on the scalp and reapply until you feel a cooling wet sensation during application - this confirms the mechanism is working and that a good amount of product is being delivered.
  Frequency: Apply the treatment twice daily- once after morning shower and once before bed time. immediately after shower and at night before bed.
  Route of administration: Topical Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Arms: Fermented Extract Hair Growth and Scalp Health Serum
Other: Placebo Hair Growth and Scalp Health Serum — Mode of Usage: Apply the serum directly to the scalp using the rollerball applicator. Gently roll the ball over thinning or affected areas of the scalp. Gently massage the serum into the scalp with clean fingertips to help it absorb fully. Ensure liquid is visible on the scalp and reapply until you feel a cooling wet sensation during application - this confirms the mechanism is working and that a good amount of product is being delivered.
  Frequency: Apply the treatment twice daily - once after morning shower and once before bed time. immediately after shower and at night before bed.
  Route of administration: Topical Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight
  Arms: Placebo Hair Growth and Scalp Health Serum

SUMMARY:
This is a Prospective, Interventional, Randomized, Double-Blind, Placebo-Controlled, Single-Centre, Clinical Study to Evaluate the Safety, Efficacy and In-Use Tolerability of Fermented Extract Hair Growth and Scalp Health Serum.

DETAILED DESCRIPTION:
A total of 34 participants, including males and non- pregnant, non-lactating females aged between 18 and 55years (inclusive) with Mild to Moderate Hair Thinning will be enrolled in the study. The study aims to complete evaluation for 30 participants, from that 20 subjects in the Treatment A group (bioactive) and 10 subjects in the Treatment B group (placebo). Scalp skin type-categorized as dry, oily, or combination-will be recorded during screening.

There will be total of 6 visits during the study. The duration of the study will be 90 Days (3 months) from the enrolment Visit 01 (Day -04, Week 00): Screening, Informed Consent, Tattoo Marking, Hair Growth Rate Visit 02 (Day 01, Week 00): Randomization, Baseline Evaluations, Buccal DNA Swab Visit 03 (Day 42, Week 06): Tattoo Marking, Hair Growth Rate Visit 04 (Day 45, Week 06): Evaluation Visit 05 (Day 87, Week 12): Tattoo Marking, Hair Growth Rate Visit 06 (Day 90, Week 12): Evaluations, Buccal DNA Swab, End of Study Evaluation parameter: Hair Growth Rate, Thickness, Density, Scalp Condition, A:T Ratio, 60 secs Hair combing, Hair Pull Test, Dermatologist Evaluation, Subjective Response Index, Global Photography of Head Crown, Graying Severity Score (GSS), Tensile Strength

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-55years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Subject is in good general health as determined by the Investigator on the basis of medical history.
5. Patients must have a confirmed diagnosis of mild to moderate hair thinning, during clinical study and grade will be evaluated by the dermatologist by using Norwood-Hamilton classification for male (Grade 1-3) and Ludwig pattern scale for female (Grade 1-2) with active hair shredding
6. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
7. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
8. Subjects are willing to give written informed consent and are willing to follow the study procedure.
9. Subjects who commit not to use any other medicated/ prescription shampoos/hair care products, any other hair growth products or hair colour or dye, other than the test treatment for the entire duration of the study.
10. Subject is willing and able to comply with study procedures, including all scheduled visits, treatment applications, and assessments.
11. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
12. Subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subject have history of severe hair fall due to any clinically significant self-reported problems like anaemia, thyroid problems.
2. Subject have history of any prior hair growth procedures done (e.g. hair transplant or laser).
3. Subject who had taken topical product of hair loss for at least 4 weeks before enrolment.
4. Subject who had taken any systemic product for any illnesses for at least 3 months.
5. History of alcohol or drug addiction.
6. Subject having history or resent condition of severely irritated or visibly inflamed scalp or severe scalp disease.
7. Subject having history or present condition of an allergic response to any cosmetic products, any other condition which could warrant exclusion from the study.
8. Pregnant or breast feeding or planning to become pregnant during the study period.
9. History of chronic illness which may influence the cutaneous state.
10. Subject have participated any clinical research study related to hair care products.
11. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or product of any type of cancer within the last 6 months.
12. Participants with advanced baldness (Norwood 4-7, Ludwig 3), long-standing bald patches (>1 year), scarring alopecia, active scalp infections, recent use of hair growth treatments (e.g., minoxidil or finasteride within the past 3 months), severe scalp conditions, or known allergies to any test product ingredients will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hair Growth Rate measured by CASLiteNova from the tattoo-marked area | Baseline (Day -4 to Day 1, prior to treatment), Day 42 (±2 days), Day 45 (±2 days), Day 87 (±2 days), and Day 90 (±2 days).
  Hair growth rate will be assessed using the CASLiteNova from the tattoo-marked area of the scalp. The change from baseline values will be compared within and across treatment arms.
Change from Baseline in Baby Hair Count and Hair Length measured by CASLiteNova from the bald scalp area | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).)
  Baby hair count and hair length will be evaluated using the CASLiteNova digital imaging system from the bald scalp area. The change from baseline values will be compared within and across treatment arms.
Change from Baseline in Hair Density and Hair Thickness measured by CASLiteNova | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  Hair density (hairs/cm²) and hair thickness (μm) will be evaluated using the CASLiteNova digital imaging system. The change from baseline values will be compared within and across treatment arms.

SECONDARY OUTCOMES:
Change from Baseline in Scalp Condition measured by CASLiteNova | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  Scalp condition will be evaluated using the CASLiteNova digital imaging system to assess improvements in scalp parameters.
Change from Baseline in Anagen-to-Telogen (A:T) Hair Ratio measured by CASLiteNova | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  The ratio of anagen to telogen hairs will be assessed using the CASLiteNova digital imaging system to evaluate hair growth phase distribution.s
Change from Baseline in Total Hair Count on the Vertex Region measured by Digital Photography and Image Pro Analysis | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  Total hair count on the vertex (crown) region of the scalp will be evaluated using standardized digital photography at a 90° angle and analyzed through image pro analysis software.
Change from Baseline in General Scalp Appearance evaluated by Dermatologist | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  General scalp appearance, including itchiness, redness, roughness, scaliness, and dryness, will be assessed by a dermatologist or a dermatologist-trained evaluator.
Improvement in general appearance of hair i.e. hair volume, hair plasticity, hair density, hair shininess, hair smoothness, hair dryness and hair strength evaluated by the Dermatologist or Dermatologist trained evaluator | Baseline (Day 01, prior to treatment usage) to post treatment assessments on Day 45 (+2 Days) and Day 90 (+2 Days)
  General hair appearance, including hair volume, plasticity, density, shininess, smoothness, dryness, and strength, will be assessed by a dermatologist or a dermatologist-trained evaluator.
Improvement in hair fall- both from the scalp root and due to hair shaft breakage evaluated through 60 second hair combing test by dermatologist trained evaluator | Baseline (Day 01, prior to treatment usage) to post treatment assessments on Day 45 (+2 Days) and Day 90 (+2 Days)
  Hair fall, including shedding from the scalp root and hair shaft breakage, will be evaluated using the 60-second hair combing test by a dermatologist-trained evaluator.
Improvement in hair root strength evaluated through hair pull test by dermatologist trained evaluator | Baseline (Day 01, prior to treatment usage) to post treatment assessments on Day 45 (+2 Days) and Day 90 (+2 Days)
  Hair root strength will be evaluated using the hair pull test by a dermatologist-trained evaluator.
Improvement in tensile strength of single hair strand evaluator through TESTRONIX tensile tester of hair | Baseline (Day 01, prior to treatment usage) to post treatment assessments on Day 45 (+2 Days) and Day 90 (+2 Days)
  Tensile strength of a single hair strand will be measured using a TESTRONIX tensile tester to assess mechanical hair strength.
Improvement in extent of hair greying as measured by a Grey Scoring Scale | Baseline (Day 01, prior to treatment usage) to post treatment assessments on Day 90 (+2 Days)
  The extent of hair greying will be assessed using a validated Grey Scoring Scale to evaluate changes from baseline.
Change from Baseline in Scalp Microbiome Composition measured by 16S rRNA Gene-Based DNA Sequencing | Baseline (Day 1, prior to treatment) and Day 90 (±2 days).
  Scalp microbiome will be assessed using BD swabs for 16S rRNA gene-based DNA sequencing to evaluate changes in microbial composition from baseline.
Change from Baseline in Treatment Perception Questionnaire Score measured by Structured Questionnaire | Baseline (Day 1, prior to treatment), Day 45 (±2 days), and Day 90 (±2 days).
  Treatment perception will be evaluated using a structured questionnaire. Scores will be compared with baseline values to assess patient-reported outcomes.
Change from Baseline in Hair Density Patterns measured by Norwood-Hamilton Scale (males) and Ludwig Scale (females) | Baseline (Day 1, prior to treatment) and Day 90 (±2 days).
  Hair density patterns will be assessed using the Norwood-Hamilton scale for male participants and the Ludwig scale for female participants. Changes from baseline will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Study Director — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No